CLINICAL TRIAL: NCT04431947
Title: Sleep and Psychosocial Outcomes After Initiation of Advanced Hybrid Closed-Loop Insulin Delivery Systems in Youth With Type 1 Diabetes and Their Parents
Brief Title: Impact of Hybrid Closed-Loop Systems on Sleep and Psychosocial Outcomes in Youth With T1D and Their Parents
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-0375; K12DK094712 (NIH)
Record Dates: First submitted 2020-06-02; First posted 2020-06-16 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Youth: Youth, between the ages of 2 and 17, with type 1 diabetes
- Parent: Parents of youth with type 1 diabetes

SUMMARY:
This study evaluates the impact of the hybrid closed-loop insulin delivery systems on sleep in youth with type 1 diabetes and their parents. Activity watches, surveys and device downloads are used to evaluate sleep in these participants.

DETAILED DESCRIPTION:
Sleep is important for everyone, including youth with type 1 diabetes. New technology has shown improvements in glycemic variability, especially overnight. This study evaluates the impact of advanced hybrid closed-loop insulin delivery systems on sleep for both youth with type 1 diabetes and their parents. Study measures include wearing an actigraphy watch and completing a sleep diary for 7 days and taking surveys on sleep and psychosocial measures. Study measures occur prior to starting the hybrid closed-loop system, immediately after starting the system and at 3 and 6 months after starting the system.

ELIGIBILITY:
Inclusion Criteria:

* Child diagnosed with type 1 diabetes for at least 3 months
* Child receives clinical care at the Barbara Davis Center for Diabetes
* Child starting an advanced HCL system as part of routine diabetes care
* Child currently living with a parent who is willing to complete surveys for this study
* Family able to read and speak English
* Parent lives at home with the child with type 1 diabetes
* Parent able to read and speak English

Exclusion Criteria:

* Child has an active underlying sleep disorder, such as narcolepsy, insomnia or untreated sleep apnea
* Child participating in an interventional research protocol
* Child unable to complete study procedures
* Parent has an active underlying sleep disorder, such as narcolepsy, insomnia or untreated sleep apnea
* Parent unable to complete study procedures

Ages: 2 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Youth with type 1 diabetes and a parent who resides with the youth.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Duration of Sleep | End of study (6 months)
  Change in duration of sleep before and after starting the advanced hybrid closed-loop system using surveys and activity watches

SECONDARY OUTCOMES:
Impact on Diabetes Distress | End of study (6 months)
  Change in diabetes-related distress using the validated Problem Areas in Diabetes survey
Impact on Quality of Life | End of study (6 months)
  Change in quality of life using the validated survey Pediatric Quality of Life Inventory Diabetes Module (PedsQL)
Impact on Fear of Hypoglycemia | End of study (6 months)
  Change in fear of hypoglycemia using the validated hypoglycemia fear survey
Impact on Perceptions of Diabetes Technology | End of study (6 months)
  Change in diabetes technology perceptions using the validated survey Diabetes Technology Questionnaire
Impact on Hybrid Closed-Loop System Use Perceptions | End of study (6 months)
  Change in perceptions of hybrid-closed loop systems using the validated INSPIRE survey
Impact of Sleep on Glycemic Variability | End of study (6 months)
  Correlation of sleep duration and glycemic variability using hybrid closed loop device download to analyze time in range, time with low glucose and time with high glucose

CONTACTS AND LOCATIONS:
Overall Officials: Erin Cobry, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Barbara Davis Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No